CLINICAL TRIAL: NCT02800291
Title: Making the Most of Mealtimes (M3): Determinants of Food Intake in Long Term Care
Brief Title: Making the Most of Mealtimes Determinants of Food Intake
Acronym: M3
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Alberta (Other); University of Manitoba (Other); Universite de Moncton (Other)
Responsible Party: Principal Investigator, Heather Keller, Research Chair, Nutrition & Aging, University of Waterloo
Other Study IDs: 20056
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Malnutrition
Keywords: food intake
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
M3 is a multi-site cross sectional study. Data were collected form 640 residents in 32 homes in Canada. The primary purpose of this study was to identify food intake in residents and compare this to recommendations, as well as determine influential determinants of food intake.

DETAILED DESCRIPTION:
This cross-sectional study has collected in-depth data at the resident, dining room, staff, and home level, focused on determinants of food intake. Dietary intake is based on three non-consecutive days of weighed and estimated food intake. Oral health and dyshphagia risk are assessed. Person directed care practices, mealtime environments and home level variables of food cost, production and delivery are ascertained.

ELIGIBILITY:
Inclusion Criteria:

* medically stable living in selected units, residing in home for more than one month consent to participate

Exclusion Criteria:

* considered end of life by staff; tube feeding

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants were residents in long term care. Eligible residents were medically stable, living in the selected units from the participating homes. They had to be reside in the home for more than 1 month and not be on tube feeding or be considered at the end of life.
Sampling Method: Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Malnutrition | 1 month
  Subjective Global Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, PhD, Principal Investigator — University of Waterloo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vucea V, Keller HH, Morrison JM, Duncan AM, Duizer LM, Carrier N, Lengyel CO, Slaughter SE. Nutritional quality of regular and pureed menus in Canadian long term care homes: an analysis of the Making the Most of Mealtimes (M3) project. BMC Nutr. 2017 Oct 23;3:80. doi: 10.1186/s40795-017-0198-3. eCollection 2017. PMID 32153857
- [Derived] Vucea V, Keller HH, Morrison JM, Duizer LM, Duncan AM, Steele CM. Prevalence and Characteristics Associated with Modified Texture Food Use in Long Term Care: An Analysis of Making the Most of Mealtimes (M3) Project. Can J Diet Pract Res. 2019 Sep 1;80(3):104-110. doi: 10.3148/cjdpr-2018-045. Epub 2019 Feb 7. PMID 30724101
- [Derived] Iuglio S, Keller H, Chaudhury H, Slaughter SE, Lengyel C, Morrison J, Boscart V, Carrier N. Construct validity of the Dining Environment Audit Protocol: a secondary data analysis of the Making Most of Mealtimes (M3) study. BMC Geriatr. 2018 Jan 22;18(1):20. doi: 10.1186/s12877-018-0708-4. PMID 29357821
- [Derived] Keller HH, Carrier N, Slaughter S, Lengyel C, Steele CM, Duizer L, Brown KS, Chaudhury H, Yoon MN, Duncan AM, Boscart VM, Heckman G, Villalon L. Making the Most of Mealtimes (M3): protocol of a multi-centre cross-sectional study of food intake and its determinants in older adults living in long term care homes. BMC Geriatr. 2017 Jan 13;17(1):15. doi: 10.1186/s12877-016-0401-4. PMID 28086754
- See also: Primary analysis results on determinants of food intake — http://dx.doi.org/10.1016/j.jamda.2017.05.003
- See also: Primary analysis results on determinants of fluid intake — http://doi.org/10.1016/j.gerinurse.2017.11.004

DOCUMENTS (1):
  • Study Protocol (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02800291/Prot_000.pdf